CLINICAL TRIAL: NCT00359190
Title: A Phase I, Open Label Study of the Safety, Pharmacokinetics and Pharmacodynamics of GW572016 in Once Daily Versus Twice Daily Dosing Regimens in Patients With Treatment- Naive Breast Cancer
Brief Title: Pharmacokinetics And Pharmacodynamics Of Lapatinib In Two Dosing Regimens In Treatment-naive Patients With Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EGF10027
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Neoplasms, Breast
Keywords: lapatinib; breast cancer; treatment-naive
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lapatinib receivers (Experimental): Subjects with treatment-naïve breast tumors will be administered lapatinib 1500 mg once daily, 1000 mg once daily, or 500 mg twice daily for a minimum of 9 days and maximum of 15 days prior to surgical resection..
  Interventions: Drug: lapatinib

INTERVENTIONS:
Drug: lapatinib — GW572016 ditosylate salt (lapatinib) will be given as 250 mg tablets via oral route

SUMMARY:
This study will examine the inhibition of ErbB1 and ErbB2 phosphorylation and downstream mediators of tumor cell growth and survival tumor tissue in treatment-naive breast cancer patients for three dosing schedules of lapatinib.

ELIGIBILITY:
Inclusion criteria:

* Clinical labs are within acceptable ranges.
* A histologically confirmed, treatment-naive, breast tumor measuring 1 cm or greater that can be readily biopsied.
* At least 18 years of age.
* Females must meet certain criteria specified in protocol.
* Ability to swallow and retain oral medication.
* Ability to follow and understand directions.

Exclusion criteria:

* Female who is pregnant or lactating.
* Medically unfit by the doctor as a result of the medical interview or physicals.
* Received treatment of an investigational drug within 4 weeks of study start.
* Currently receiving treatment with prohibited meds listed in protocol.
* Had major surgery in previous 2 weeks.
* Had prior radiation therapy to the chest to treat this incidence of breast cancer.
* Hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study med.
* Has a malabsorption syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2004-06-29 (Actual); Primary Completion 2008-01-09 (Actual); Study Completion 2008-01-09 (Actual)

PRIMARY OUTCOMES:
Comparison of the effects of 3 dosing schedules of lapatinib on biomarkers involved in regulating tumor cell proliferation and survival in pre-treatment and post-treatment breast tumor tissue samples. | subjects on study up to 15 days
  biomarker analysis of tumor biopsies pre/post dose

SECONDARY OUTCOMES:
Evaluation of adverse events and changes in lab values from pre-dose and post-dose. Assessment of safety & tolerability of lapatinib at multiple doses when administered to patients who have not have not been treated for breast tumors. | subjects on study up to 15 days
  safety assessments of labs, hematology labs, Electrocardiogram, vital signs

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- United States (8):
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Allentown, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Roanoke, Virginia
  - GSK Investigational Site, Milwaukee, Wisconsin
- Israel (2):
  - GSK Investigational Site, Ramat Gan
  - GSK Investigational Site, Zrifin

REFERENCES:
- [Derived] Spector NL, Robertson FC, Bacus S, Blackwell K, Smith DA, Glenn K, Cartee L, Harris J, Kimbrough CL, Gittelman M, Avisar E, Beitsch P, Koch KM. Lapatinib Plasma and Tumor Concentrations and Effects on HER Receptor Phosphorylation in Tumor. PLoS One. 2015 Nov 16;10(11):e0142845. doi: 10.1371/journal.pone.0142845. eCollection 2015. PMID 26571496
- See also: Results for study EGF10027 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/EGF10027?search=study&search_terms=EGF10027#rs